CLINICAL TRIAL: NCT06026410
Title: Phase 1, First-in-Human, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of KO-2806 When Administered as Monotherapy and in Combination Therapy in Adult Patients With Advanced Solid Tumors
Brief Title: KO-2806 Monotherapy and Combination Therapies in Advanced Solid Tumors
Acronym: FIT-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KO-2806-001
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors With HRAS Alterations; Non Small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma (PDAC); Clear Cell Renal Cell Carcinoma (ccRCC); Renal Cell Carcinoma (Kidney Cancer); Non Clear Cell Renal Cell Carcinoma (nccRCC)
Keywords: HRAS; KRAS; NRAS; Farnesyltransferase inhibitor (FTI); Tyrosine Kinase inhibitor (TKI); Phase 1; KRAS G12C inhibitor; NSCLC; ccRCC; RCC; PDAC; CRC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms | interventions — cabozantinib; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm #1: RAS-altered advanced solid tumors, monotherapy (escalation phase) (Experimental): Patients with advanced solid tumors and the following:
  * HRAS-mutant and/or amplified tumors (any solid tumor type)
  * HRAS overexpression (only for HNSCC tumors)
  * KRAS and/or NRAS and/or HRAS-mutant and/or amplified for NSCLC or CRC
  * KRAS-mutant and/or amplified PDAC
  Interventions: Drug: Darlifarnib
- Arm #2: Advanced or metastatic RCC, combination therapy (escalation phase) (Experimental): Patients who have received at least 1 prior systemic therapy with immuno-oncology (IO)-based treatment for locally advanced or metastatic RCC with predominantly clear cell subtype; non-clear cell RCC patients who are either treatment naïve or have received any prior systemic treatment for locally advanced and metastatic RCC
  Interventions: Drug: Darlifarnib; Drug: Cabozantinib
- Arm #3: Advanced or metastatic NSCLC, CRC, or PDAC, combination therapy (escalation phase) (Experimental): Patients with KRAS G12C-mutant locally advanced or metastatic NSCLC, CRC, or PDAC who have received at least 1 prior systemic therapy including available approved standard of care treatments
  Interventions: Drug: Darlifarnib; Drug: Adagrasib
- Arm #4: Advanced or metastatic ccRCC, combination therapy (expansion phase) (Experimental): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC
  Interventions: Drug: Darlifarnib; Drug: Cabozantinib
- Arm #5: Advanced or metastatic ccRCC, monotherapy (expansion phase) (Experimental): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC
  Interventions: Drug: Cabozantinib
- Arm #6: Advanced or metastatic ccRCC, cabozantinib rollover to combination therapy (expansion phase) (Experimental): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC
  Interventions: Drug: Darlifarnib; Drug: Cabozantinib
- Arm #7: Advanced or metastatic NSCLC, combination therapy (expansion phase) (Experimental): Patients with KRAS G12C-mutant locally advanced or metastatic NSCLC who have received at least 1 prior systemic therapy including available approved standard of care treatments
  Interventions: Drug: Darlifarnib; Drug: Adagrasib

INTERVENTIONS:
Drug: Darlifarnib — Oral administration
  Other Names: KO-2806
  Arms: Arm #1: RAS-altered advanced solid tumors, monotherapy (escalation phase); Arm #2: Advanced or metastatic RCC, combination therapy (escalation phase); Arm #3: Advanced or metastatic NSCLC, CRC, or PDAC, combination therapy (escalation phase); Arm #4: Advanced or metastatic ccRCC, combination therapy (expansion phase); Arm #6: Advanced or metastatic ccRCC, cabozantinib rollover to combination therapy (expansion phase); Arm #7: Advanced or metastatic NSCLC, combination therapy (expansion phase)
Drug: Cabozantinib — Oral administration
  Other Names: Cabometyx
  Arms: Arm #2: Advanced or metastatic RCC, combination therapy (escalation phase); Arm #4: Advanced or metastatic ccRCC, combination therapy (expansion phase); Arm #5: Advanced or metastatic ccRCC, monotherapy (expansion phase); Arm #6: Advanced or metastatic ccRCC, cabozantinib rollover to combination therapy (expansion phase)
Drug: Adagrasib — Oral administration
  Other Names: Krazati
  Arms: Arm #3: Advanced or metastatic NSCLC, CRC, or PDAC, combination therapy (escalation phase); Arm #7: Advanced or metastatic NSCLC, combination therapy (expansion phase)

SUMMARY:
This first-in-human (FIH) dose-escalation and dose-validation/expansion study will assess KO-2806, a farnesyltransferase inhibitor (FTI), as a monotherapy and in combination, in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Histologically or cytologically confirmed advanced solid tumors

  * Arm #1 (KO-2806 monotherapy): Patients who have progressed on, or are refractory to, standard of care (SOC) treatments with advanced solid tumors, specifically: HRAS-mutant and/or amplified tumors (any solid tumor type); HRAS overexpression (only for HNSCC tumors); KRAS and/or NRAS, and/or HRAS-mutant and/or amplified NSCLC or CRC; KRAS-mutant and/or amplified PDAC
  * Arm #2 (Combination): Patients who have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic RCC with predominantly clear cell subtype; non-clear cell RCC patients who are either treatment-naïve or have received any prior systemic treatment for locally advanced and metastatic RCC.
  * Arm #3 (Combination): Patients who have received at least 1 prior systemic therapy including available approved SOC treatments for KRAS G12C-mutant locally advanced or metastatic NSCLC, CRC, or PDAC.
  * Arm #4 (Combination): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC, but no more than 3 prior systemic anticancer therapies.
  * Arm #5 (Cabozantinib monotherapy): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC, but no more than 3 prior systemic anticancer therapies.
  * Arm #6 (Cabozantinib rollover to combination): Patients must be cabozantinib-naïve and have received at least 1 prior systemic therapy with IO-based treatment for locally advanced or metastatic ccRCC, but no more than 3 prior systemic anticancer therapies.
  * Arm #7 (Combination): Patients who have received at least 1 prior systemic therapy including available approved SOC treatments for KRAS G12C-mutant locally advanced or metastatic NSCLC
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Karnofsky Performance Status of 70 or higher with no clinically significant deterioration over the previous 2 weeks.
* Acceptable liver, renal, endocrine, and hematologic function.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any use of anticancer therapy within 14 days or 5 half-lives (whichever is shorter) of Cycle 1 Day 1.
* Prior treatment with an FTI or HRAS inhibitor.
* Major surgery, other than local procedures, within 28 days prior to Cycle 1 Day 1, without complete recovery.
* Spinal cord compression, leptomeningeal disease, or clinically active CNS metastases.
* Toxicity (excluding alopecia) from prior therapy that has not been completely resolved to baseline at the time of consent.
* Active or prior documented autoimmune or inflammatory disorders within the past 5 years prior to Cycle 1 Day 1 (with exceptions).
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
* Inability to swallow, impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the trial drugs.
* Inadequate cardiac and/or vascular function, including receipt of treatment for unstable angina, myocardial infarction, and/or cerebrovascular attack within the prior 6 months, mean QTcF ≥470 ms, or Class II or greater congestive heart failure.
* Other invasive malignancy within 2 years.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) | DLTs will be evaluated during the first 28 days of KO-2806 treatment (dose escalation)
Descriptive statistics of adverse events (AEs) | First dose of KO-2806 up to and including 28 days after last dose of KO-2806 (dose escalation)
  NCI-CTCAE v5.0
Incidence of dose interruptions, reductions, and discontinuations due to AE | First dose of KO-2806 up to last dose of KO-2806 or up to 24 months of treatment (dose escalation)
Objective Response Rate (ORR) | Up to an estimated period of 24 months (dose expansion)
  Assessed per RECIST v1.1

SECONDARY OUTCOMES:
Incidence of dose interruptions, reductions, and discontinuations due to AE | First dose of KO-2806 up to last dose of KO-2806 or up to 24 months of treatment (dose expansion)
Descriptive statistics of AEs | First dose of KO-2806 up to and including 28 days after last dose of KO-2806 (dose expansion)
  NCI-CTCAE v5.0
Objective Response Rate (ORR) | Up to an estimated period of 24 months (dose escalation)
  Assessed per RECIST v1.1
Disease control rate (DCR) | Up to an estimated period of 24 months (dose escalation and expansion)
  Assessed per RECIST v1.1
Duration of response (DoR) | Up to an estimated period of 24 months (dose escalation and expansion)
  Assessed per RECIST v1.1
Time to response (TTR) | Up to an estimated period of 24 months (dose escalation and expansion)
  Assessed per RECIST v1.1
Progression-Free Survival (PFS) | Up to an estimated period of 24 months (dose escalation and expansion)
  Assessed per RECIST v1.1
Overall Survival (OS) | First dose of KO-2806 until death, or up to an estimated period of 37 months (dose escalation and expansion)
  For patients with no events, OS will be censored at the last known to be alive date
AUClast | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Area under the curve from time zero to last measurable concentration for KO-2806 (in the absence and presence of food) and combination agent.
AUC0-inf | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Area under the curve from time zero to infinity post administration for KO-2806 (in the absence and presence of food) and combination agent
Cmax | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Maximum plasma concentration (Cmax) of KO-2806 (in the absence and presence of food) and the combination agent
Cmin | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Minimum plasma concentration (Cmin) of KO-2806 (in the absence and presence of food) and the combination agent
Tmax | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Time to maximal concentration (Tmax) of KO-2806 (in the absence and presence of food) and the combination agent
Estimated terminal elimination rate constant (λz) | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Estimated terminal elimination rate constant of KO-2806 and the combination agent
t1/2 | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Half-life (t1/2) of KO-2806 (in the absence and presence of food) and the combination agent
CL/F | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Total apparent clearance (CL/F) of KO-2806 and the combination agent
Vd/F | Cycle 1. Each cycle is 28 days. (Dose escalation and dose expansion)
  Total apparent volume of distribution (Vd/F) of KO-2806 and the combination agent
QTcF | Up to 28 days following last dose of KO-2806, cabozantinib, or adagrasib. (Dose escalation and dose expansion)
  QT interval corrected for heart rate (HR) using Fridericia's formula (QTcF) for KO-2806 monotherapy and in combination
KO-2806 plasma concentration measurements | Up to day 28 following first dose of KO-2806 and adagrasib. (Dose escalation and dose expansion)
Amount of KO-2806 excretion in urine | Up to 24 hours following first dose of KO-2806. (Dose escalation)
CLr of KO-2806 excretion in urine | Up to 24 hours following first dose of KO-2806. (Dose escalation)
  Renal clearance of KO-2806 excretion in urine

CONTACTS AND LOCATIONS:
Locations (32):
- United States (20):
  - Mayo Clinic Comprehensive Cancer Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Department of Medicine, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - AdventHealth Celebration, Celebration, Florida
  - Mayo Clinic Comprehensive Cancer Center, Jacksonville, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Comprehensive Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - OU Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI - Oncology Partners, Nashville, Tennessee
  - UT Southwestern Simmons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin (Carbone Cancer Center), Madison, Wisconsin
- France (3):
  - Oncologie médicale - Pitié-Salpêtrière, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Fondazione Piemonte per l'Oncologia - IRCCs Candiolo, Candiolo
  - Istituto Nazionale Tumori IRCCS, Napoli
  - Camplus Humanitas University, Rozzano
  - AOU Verona - Centro Ricerche Cliniche di Verona, Verona
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital HM Sanchinarro START Madrid-CIOCC, Madrid
  - Hospital Universitario Virgen del Rocío, Seville